CLINICAL TRIAL: NCT03759054
Title: Cancer Patients in Clinical Trials and Their Relatives
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulrik Lassen, Head of Department of Oncology, professor, Rigshospitalet, Denmark
Other Study IDs: Fase 1 patienter
Record Dates: First submitted 2017-05-05; First posted 2018-11-29 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Depression, Anxiety; Information Disclosure
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aims

The aims of this study are:

1. To characterize patients' psychological well-being from the time they are referred to a phase I trial and determine risk factors for poor well-being.
2. To investigate perceived information, expectations and regret when a patient participate in a phase I trial.

Materials and methods This study is a prospective cohort study based on longitudinal applied questionnaires.

The questionnaire will consist of questionnaires measuring stress, anxiety, depression and health-related quality of life longitudinal through the course in the Phase I Unit. At the time of inclusion in a trial, there will be questions regarding perceived information and expectations. At the time of exclusion from trial, there will be questions regarding regret.

The questionnaire will consist primarily of validated questionnaires. When a validated questionnaire does not exist, a previous applied questionnaire will be used to ensure comparison with data from other studies. Only a limited use of self-constructed single-items will be applied.

DETAILED DESCRIPTION:
Background The association between cancer and the occurrence of psychological disturbances has been shown in several studies. For cancer patients participating in phase I trials, psychological disturbances have also been found to be present, although with no comparison group.

Relatives to patients in phase I trials are also found to have higher levels of perceived stress and anxiety among 88 relatives compared to population norms measured with validated instruments.

Recognizing the aim of a phase I trial as dose escalation was found among a minority of patients (mean, 33%; range, 17-44%) in a systematic review. This review also found that a mean of 62% (range, 22-92%) of patients expected personal benefit from the new drug and a mean of 27% (range, 7-38%) expecting a cure for their cancer.

Regret has only been explored to a limited extent among patients in phase I trials and has only been found among a minority.

Applied scales in the study

* Psychological well-being will be measured with the Perceived Stress Scale (PSS), the Generalized Anxiety Disorder (GAD7), and the Patient Health Questionnaire (PHQ-9).
* Health-related quality of life will be measured with the EORTC Quality of Life Questionnaire (QLQ-C30) for patients and the Short-Form Health Survey (SF-36) for relatives.
* Quality of Informed Consent (QuIC)
* Expectations
* Decision Regret Scale

Perspectives This study will contribute with a characterization of the psychological well-being of patients referred to the Phase I Unit and possible factors of importance for this, including the relatives' well-being. This knowledge can lead to a greater attention to patients at risk of developing psychological disturbances and define challenges for recruitment and maintenance in phase I trials.

The study will contribute to knowledge of patients' understanding of phase I trials and how this can affect expectations and regret. Moreover, this study will be the first to investigate if relatives' understanding of trial influences patients' perception of trial. These findings are important for the evaluation the dialogue when information is given and to considerations regarding involvement of relatives as possible resources for the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the Phase I Unit

Exclusion Criteria:

* patients who do not understand written Danish
* patients for whom contact information is missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and referred to the Phase I Unit at the Department of Oncology, Rigshospitalet, and their closest relative will be invited to participate when they come for their first information dialogue in the department. The questionnaire can be filled out immediately after the dialogue if possible or filled out at home and sent or brought to the department at next appointment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Stress assessed by the Perceived Stress Scale, total score (range 0-40), higher score indicates a higher level of stress. | First visit, at baseline visit, day 42 visit, through study completion, an average of 1 year
  Among patients and relatives
Anixiety assessed by Generalized Anxiety Disorder scale, total score (range 0-21), higher score indicates a higher level of anxiety. | First visit, at baseline visit, day 42 visit, through study completion, an average of 1 year
  Among patients and relatives
Depression assessed by Patient Health Questionnaire, total score (range 0-28), higher scoreindicates a higher level of depression. | First visit, at baseline visit, day 42 visit, through study completion, an average of 1 year
  Among patients and relatives
Physical functioning assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, subscale physical functioning, score (range 0-100), higher score indicates better physical functioning. | First visit, through study completion, an average of 1 year
  Patients

SECONDARY OUTCOMES:
Perceived information assessed by the QuIC, total score (range 0-100), higher score indicates a higher level of knowledge | At baseline visit
  Among patients and relatives
Regret assessed by Decision Regret Scale, total score (range 0-100), higher score indicates higher level of regret | through study completion, an average of 1 year
  Among patients only
Question regarding motivations: How did you get to hear about the Phase 1 Unit? Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding motivations: Indicate your reasons for participating in clinical trial treatment by circling the relevant number. Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding expectations: During the clinical trial treatment do you expect your tumour(s) to … ? Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding expectations: Do you expect the side effects of the clinical trial treatment to be … ? Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding expectations: If you have received chemo treatment previously, how do you expect the side effects of the clinical trial treatment will be? Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding expectations: Would you like to participate in a phase 1 trial? Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding expectations: Does your family or do your friends want you to participate in a phase 1 trial? Descriptive distribution of answers. | At baseline visit
  Among patients only
Question regarding expectations: I expect: That my physically health will improve/That my mental health will improve/That my life from a social aspect will improve/That I will prolong my life/That I will be cured. Descriptive distribution of answers. | At baseline visit
  Among patients only

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD, Study Director — Head of Department of Oncology
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No